CLINICAL TRIAL: NCT04866732
Title: Physical Activity Program for Cardiac Health Among Older African American Populations Living in Rural Alabama: Needs Assessment and Initial Development
Brief Title: Physical Activity Program for Cardiac Health Among Older African American Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 000526161
Record Dates: First submitted 2021-04-20; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Cardiovascular; Disease
Keywords: Cardiovascular; African American; Older; Women; Rural
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: This project involves a mixed methods study with sequential design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Needs assessment and feasibility group (Experimental): Based on our target population's needs/preferences, an existing Physical Activity (PA) program will be modified and tailored to the needs of the target population. We anticipate that this PA program will include the following components: a) PA component - ( duration of walk) from baseline to the end of the study; b) weekly informational sessions on various topics related to CVD risk factors prevention; c) daily diary to record if they are facing any barriers in completing various components of the intervention; d) problem-solving sessions
  Interventions: Behavioral: Physical Activity Cardiac Health Program

INTERVENTIONS:
Behavioral: Physical Activity Cardiac Health Program — The investigators anticipate that the physical activity program will include the following components: a) physical activity component - the investigators propose an incremental physical activity component whereby participants will gradually increase their physical activity ( duration of walk) from baseline to the end of the study; b) weekly informational sessions on various topics related to Cardiovascular disease risk factors prevention; c) daily diary, which will be used to document record about any barriers for completing various components of the intervention; d) problem-solving sessions whereby participants will meet once a week with the investigators to talk about the barriers and facilitators of their weekly activity and any adherence issues.

SUMMARY:
Cardiovascular Diseases (CVD) are the leading cause of morbidity and mortality globally, and older African Americans (AAs) living in rural areas are disproportionately affected by this healthcare problem. The investigators propose conducting a mixed-methods study to gain information about CVD-related knowledge, perceptions regarding CVD-related healthcare needs, preferences and access barriers, and cultural aspects within this population. The information will be used in tailoring an existing intervention to meet those needs and preferences and evaluate its feasibility among older AAs living in rural Alabama. This study will lay a foundation for developing a federal grant application and a line of independent research by this early-stage investigator.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) are a leading cause of morbidity and mortality. Older populations are inherently more vulnerable to such conditions. Older African American (AA) populations living in rural areas are disproportionately affected by CVD, which has been shown to cause an increased risk for mortality in this population. Evidence suggests using lifestyle Physical activity programs to prevent CVD risk factors, which can decrease the morbidity and mortality rates associated with these health conditions. There are limited resources and healthcare services available to these populations, especially those living in Alabama's black belt. Therefore, this research project proposes conducting a phased mixed-methods study to collect data from rural AA older adults. These data are the critical first step towards developing a culturally sensitive, accessible, and acceptable intervention that addresses their needs and risk factors, incorporates their preferences, and mitigates identified barriers, which will be tested for feasibility and acceptability in this pilot study. The aims for this study are Aim 1: Through survey and interviews, assess: i) the knowledge and perceptions of AA older adults living in rural Alabama regarding CVD-related risk factors; ii) the needs/existing resources and access barriers for a community-based physical activity program; iii) the perceptions about a proposed intervention and its components, method of delivery, time/effort, and incentives; and iv) the cultural preferences regarding recruitment strategies, treatment strategies, and incentives. Aim2a: Based on the findings of Aim 1, develop a PA program for improving CVD-related risk factors among older AA populations living in rural Alabama. Aim2b: To examine the feasibility and acceptability of delivering a PA program (developed in Aim 2a) among the older AA populations living in rural Alabama. The enhanced program would enable AA older populations to prevent and manage CVD-related risk factors. It will also help in filling the gap of health disparity between AAs and other ethnicities.

ELIGIBILITY:
Inclusion Criteria:

* AA women above 65 years of age
* residing in a community setting of rural Alabama
* diagnosis of CVD
* two or more CVD-related risk factors
* able to speak and understand English
* physically inactive (engaging in no structured ambulatory/walking based lifestyle physical activity),
* able to understand and participate in basic elements (informed consent, components of intervention) of the study.

Exclusion Criteria:

* medical co-morbidity or any acute illness or frailty that would prevent their participation in the physical activity component,
* history of more than two falls in the last two months
* suicidal ideation
* scoring below 22 on Mini-Mental Status Examination Scale
* lack of transportation to the research sites
* concurrent participation in any other heart health or Physical activity intervention study.
* engaged in any kind of ambulatory/walking-based lifestyle physical activity

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Only those participants who identify themselves as female gender will be recruited.
Enrollment: 30 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Physical Activity | 12 Weeks
  The investigators will measure the leisure-time physical activity including walk. This will be measured by an accelerometer which gives more accurate information about the ambulation of a person. Scores can range between 0 and infinite.
  The higher the score, the better is the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mudasir Andrabi, Ph D, Principal Investigator — The University of Alabama; Robert Motl, Ph D, Study Director — The University of Alabama at Birmingham; Karlene Ball, Ph D, Study Director — The University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: Yes
The investigators expect that the results of the proposed study will be of great interest to the scientific community. Investigators will collect and analyze the data for the course of the study and allow one calendar year from the end of the budget period to complete data analysis and publication of results. In the interim, data will be presented at scientific meetings and shared with providers and clinicians, surrounding prevention and treatment centers, and appropriate councils and organizations, such as the Alabama Department of Public Health and academic institutions with a curriculum focused on Cardiovascular disease prevention education. The findings will be disseminated using peer-reviewed journals and presentations at local, national, and international conferences. All these avenues are instrumental in the successful dissemination of the research findings. The investigators will also ensure that the NIA has access to our data through clinicaltrials.gov.
Supporting Information: CSR
Time Frame: Immediately following publication- 36 months following publication
Access Criteria: Anyone who wish to access the data.

REFERENCES:
- [Result] Abbott LS, Slate EH. Improving Cardiovascular Disease Knowledge among Rural Participants: The Results of a Cluster Randomized Trial. Healthcare (Basel). 2018 Jun 25;6(3):71. doi: 10.3390/healthcare6030071. PMID 29941776
- [Result] Abu Alhaija ES, Aldaikki A, Al-Omairi MK, Al-Khateeb SN. The relationship between personality traits, pain perception and attitude toward orthodontic treatment. Angle Orthod. 2010 Nov;80(6):1141-9. doi: 10.2319/012710-59.1. PMID 20677967
- [Result] Agrell B, Dehlin O. Comparison of six depression rating scales in geriatric stroke patients. Stroke. 1989 Sep;20(9):1190-4. doi: 10.1161/01.str.20.9.1190. PMID 2772980
- [Result] Andrawes WF, Bussy C, Belmin J. Prevention of cardiovascular events in elderly people. Drugs Aging. 2005;22(10):859-76. doi: 10.2165/00002512-200522100-00005. PMID 16245959
- [Result] Angermayr L, Melchart D, Linde K. Multifactorial lifestyle interventions in the primary and secondary prevention of cardiovascular disease and type 2 diabetes mellitus--a systematic review of randomized controlled trials. Ann Behav Med. 2010 Aug;40(1):49-64. doi: 10.1007/s12160-010-9206-4. PMID 20652464
- [Result] Bellet RN, Adams L, Morris NR. The 6-minute walk test in outpatient cardiac rehabilitation: validity, reliability and responsiveness--a systematic review. Physiotherapy. 2012 Dec;98(4):277-86. doi: 10.1016/j.physio.2011.11.003. Epub 2012 May 16. PMID 23122432
- [Result] Cho D, Nguyen NT, Strong LL, Wu IHC, John JC, Escoto KH, Wetter DW, McNeill LH. Multiple Health Behaviors Engagement in an African American Cohort: Clustering Patterns and Correlates. Health Educ Behav. 2019 Jun;46(3):506-516. doi: 10.1177/1090198119826207. Epub 2019 Feb 18. PMID 30776919
- [Result] Colantonio LD, Monda KL, Rosenson RS, Brown TM, Mues KE, Howard G, Safford MM, Yedigarova L, Farkouh ME, Muntner P. Characteristics and Cardiovascular Disease Event Rates among African Americans and Whites Who Meet the Further Cardiovascular Outcomes Research with PCSK9 Inhibition in Subjects with Elevated Risk (FOURIER) Trial Inclusion Criteria. Cardiovasc Drugs Ther. 2019 Apr;33(2):189-199. doi: 10.1007/s10557-019-06864-2. PMID 30746585
- [Result] Der Ananian C, Winham DM, Thompson SV, Tisue ME. Perceptions of Heart-Healthy Behaviors among African American Adults: A Mixed Methods Study. Int J Environ Res Public Health. 2018 Nov 1;15(11):2433. doi: 10.3390/ijerph15112433. PMID 30388803
- [Result] Ferdinand DP, Nedunchezhian S, Ferdinand KC. Hypertension in African Americans: Advances in community outreach and public health approaches. Prog Cardiovasc Dis. 2020 Jan-Feb;63(1):40-45. doi: 10.1016/j.pcad.2019.12.005. Epub 2019 Dec 19. PMID 31863786
- [Result] Garatachea N, Torres Luque G, Gonzalez Gallego J. Physical activity and energy expenditure measurements using accelerometers in older adults. Nutr Hosp. 2010 Mar-Apr;25(2):224-30. PMID 20449530